CLINICAL TRIAL: NCT04711551
Title: Patients-reported Outcome Measures (PROMs), Clinical Objective and Biomolecular Assessment for the Monitoring of Patients Undergoing Regenerative Medicine Treatments with Orthobiologics
Brief Title: Clinical and Biomolecular Assessment for the Monitoring of Patients Undergoing Regenerative Medicine Treatments with Orthobiologics
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: REGAIN
Record Dates: First submitted 2020-12-23; First posted 2021-01-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal System Disease
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Combination Product: PRP and related devices to abtain platelet concentrate from whole blood, medullary and adipose tissue and related devices — PRP and related devices to abtain platelet concentrate from whole blood, medullary and adipose tissue and related devices

SUMMARY:
the aim is to improve the evaluation of the outcomes of regenerative medicine treatments performed in the regenerative medicine centers involved in the study.

patients who undergo regenerative medicine treatments present acute and chronic pathologies of the musculoskeletal system, of the stomatological system and of the integuments.

Objective pre, peri and post treatment evaluations are collected. A dedicated software collects the PROMs compiled by the patients, the objective clinical data and the biomolecular evaluations.

ELIGIBILITY:
Inclusion Criteria:

* patients who received indication for regerative medicine treatment for one of the following pathologies: Knee or hip or ankle osteoarthritis, patellar or Achilles tendon pain, shouder or elbow pain;
* males and females;
* age >= 6 years.

Exclusion Criteria:

* age < 6 years
* patients not compliant with post-treatment monitoring procedures
* pregnancy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who received indication for regerative medicine treatment for one of the following pathologies: Knee or hip or ankle osteoarthritis, patellar or Achilles tendon pain, shouder or elbow pain;
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Change between baseline and 12 months
  Pain will be measured with Visual Analog Scale (0-10, where 0 rapresents absence of pain and 10 the maximum pain possible) before and after treatment.

SECONDARY OUTCOMES:
Change in Tegner Activity Scale | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Level of activity will be recorded using Tegner activity scale (0-10, where 0 represents absence of physical activity and 10 represents national level sport activity) before and after treatment
Change in Knee injury and Osteoarthritis Outcome Score for patients affected by knee osteoarthritis | Changes between baseline and 2-, 6- 12 and 24-month assessments
  The level of symptoms, pain, activity, sport and quality of life will be assessed using Knee injury and Osteoarthritis Outcome Score (0-100, where 0 represents the worst outcome and 100 the best outcome) before and after treatment.
Change in Hip injury and Osteoarthritis Outcome Score for patients affected by hip osteoarthritis | Changes between baseline and 2-, 6- 12 and 24-month assessments
  The level of symptoms, pain, activity, sport and quality of life will be assessed using Hip injury and Osteoarthritis Outcome Score (0-100, where 0 represents the worst condition and 100 the best condition) before and after treatment.
Change in QuickDASH (Disabilities of the Arm, Shoulder and Hand) and SPADI (Shoulder Pain and Disability Index ) questionnaire for patients affected by shoulder disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  The level of symptoms, pain, activity, sport and quality of life will be assessed using Hip injury and Osteoarthritis Outcome Score (0-100, where 0 represents the worst condition and 100 the best condition) before and after treatment.
Change in the Shoulder Pain and Disability Index (SPADI) for patients affected by shoulder disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Pain level and extent of difficulty with the activity of daily living will be assessed using SPADI (0-100, where 100 represents the worst condition and 0 the best condition) in patients affected by shoulder disorders.
Change in Victorian Institute of Sport Assessment for Patellar tendon (VISA-P) score for patients affected by patellar tendon disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Symptoms, ability to perform daily and sport activities will be measured using VISA-P score (0-100, where 0 represents the worst condition and 100 the best condition) in patients affected by patellar tendon disorders.
Change in Lysholm Knee Score for patients affected by patellar tendon disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Lysholm knee score will be used to assess the condition of the knee in patients affected by patellar tendon disorders (0-100, where 0 represents the worst condition and 100 the best condition).
Change in Foot Function Index (FFI) for patients affected by ankle and foot disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Pain, Disability, and Activity Limitation in patients affected by foot and ankle disorders will be measured using FFI (0-100, where 100 represents the worst condition and 0 the best condition).
Change in Victorian Institute of Sport Assessment for Achilles tendon (VISA-A) score for patients affected by Achilles tendon disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Symptoms, ability to perform daily and sport activities will be measured in patients affected by Achilles tendon disorders using VISA-A score (0-100, where 0 represents the worst condition and 100 the best condition).
Change in Patient-Rated Tennis Elbow Evaluation (PRTEE) scale for patients affected by elbow disorders | Changes between baseline and 2-, 6- 12 and 24-month assessments
  Pain and function will be measured in patients affected by elbow disorders using PRTEE score (0-100, where 100 represents the worst condition and 0 the best condition).
Platelet count in Platelet-rich Plasma (PRP) | Baseline only
  For each patient receiving PRP, platelet count will be measured in order to evaluate possible correlation between the product composition and the clinical outcomes
Nucleated cell counts in adipose tissue- and bone marrow-derived orthobiologics | Baseline only
  For each patient receiving adipose tissue- or bone marrow-derived orthobiologics, the number of nucleated cells will be determined to evaluate possible correlation between the product composition and the clinical outcomes
Change in Visual Analog Scale | Changes between baseline and 2-, 6- and 24-month assessments
  Pain will be measured with Visual Analog Scale (0-10, where 0 rapresents absence of pain and 10 the maximum pain possible) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura De Girolamo, Principal Investigator — I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Locations (2):
- Italy (2):
  - Istituto Clinico San Siro (satellite center), Milan, Italia
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio (coordinator), Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzocca AD, McCarthy MB, Chowaniec DM, Dugdale EM, Hansen D, Cote MP, Bradley JP, Romeo AA, Arciero RA, Beitzel K. The positive effects of different platelet-rich plasma methods on human muscle, bone, and tendon cells. Am J Sports Med. 2012 Aug;40(8):1742-9. doi: 10.1177/0363546512452713. Epub 2012 Jul 16. PMID 22802273
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] Kern S, Eichler H, Stoeve J, Kluter H, Bieback K. Comparative analysis of mesenchymal stem cells from bone marrow, umbilical cord blood, or adipose tissue. Stem Cells. 2006 May;24(5):1294-301. doi: 10.1634/stemcells.2005-0342. Epub 2006 Jan 12. PMID 16410387
- [Background] Strioga M, Viswanathan S, Darinskas A, Slaby O, Michalek J. Same or not the same? Comparison of adipose tissue-derived versus bone marrow-derived mesenchymal stem and stromal cells. Stem Cells Dev. 2012 Sep 20;21(14):2724-52. doi: 10.1089/scd.2011.0722. Epub 2012 May 9. PMID 22468918
- [Background] Vishnubalaji R, Al-Nbaheen M, Kadalmani B, Aldahmash A, Ramesh T. Comparative investigation of the differentiation capability of bone-marrow- and adipose-derived mesenchymal stem cells by qualitative and quantitative analysis. Cell Tissue Res. 2012 Feb;347(2):419-27. doi: 10.1007/s00441-011-1306-3. PMID 22287041
- [Background] Caplan AI, Correa D. The MSC: an injury drugstore. Cell Stem Cell. 2011 Jul 8;9(1):11-5. doi: 10.1016/j.stem.2011.06.008. PMID 21726829
- [Background] Bosetti M, Borrone A, Follenzi A, Messaggio F, Tremolada C, Cannas M. Human Lipoaspirate as Autologous Injectable Active Scaffold for One-Step Repair of Cartilage Defects. Cell Transplant. 2016;25(6):1043-56. doi: 10.3727/096368915X689514. Epub 2015 Sep 21. PMID 26395761
- [Background] Pak J, Lee JH, Park KS, Jeong BC, Lee SH. Regeneration of Cartilage in Human Knee Osteoarthritis with Autologous Adipose Tissue-Derived Stem Cells and Autologous Extracellular Matrix. Biores Open Access. 2016 Aug 1;5(1):192-200. doi: 10.1089/biores.2016.0024. eCollection 2016. PMID 27588219
- [Background] Moatshe G, Morris ER, Cinque ME, Pascual-Garrido C, Chahla J, Engebretsen L, Laprade RF. Biological treatment of the knee with platelet-rich plasma or bone marrow aspirate concentrates. Acta Orthop. 2017 Dec;88(6):670-674. doi: 10.1080/17453674.2017.1368899. Epub 2017 Aug 23. PMID 28831830
- [Background] Centeno C, Pitts J, Al-Sayegh H, Freeman M. Efficacy of autologous bone marrow concentrate for knee osteoarthritis with and without adipose graft. Biomed Res Int. 2014;2014:370621. doi: 10.1155/2014/370621. Epub 2014 Sep 7. PMID 25276781